CLINICAL TRIAL: NCT00803621
Title: Cerebral Toxoplasmosis and AIDS in the French Departments of America (DFA). Diagnostic Contribution of a PCR Assay and Genetic Diversity of Toxoplasma Gondii.
Brief Title: Cerebral Toxoplasmosis and AIDS
Acronym: TOXODFA
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I07009
Record Dates: First submitted 2008-12-02; First posted 2008-12-05 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2013-12

CONDITIONS: Cerebral Toxoplasmosis; AIDS
MeSH Terms: conditions — Toxoplasmosis, Cerebral; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Toxoplasma PCR assay — Toxoplasma PCR assay

SUMMARY:
With a HIV incidence much higher in the DFA than in European French territory, this disease is a major public health problem in these areas, especially in French Guiana.

Cerebral toxoplasmosis is a priority among the opportunistic infections in AIDS patients from the DFA because of its frequency (French West Indies) and of its lethality (French Guiana).

The diagnosis of cerebral toxoplasmosis may be difficult because based only on presumptive clinical and radiological features. The response to specific antitoxoplasmic therapy confirms a posteriori the diagnosis.

In reference to the data collected by the Biological Resource Centre Toxoplasma, in particular in French Guiana, we think that T. gondii strains reactivating in AIDS patients from DFA are genetically different from those reactivating in AIDS patients from Europe, with an increased capacity for dissemination via peripheral blood in the first ones. This more frequent or more prolonged parasitemia could facilitate the diagnosis of cerebral toxoplasmosis by PCR test from peripheral blood samples in AIDS patients from the French departments of America.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 18 years)
* Patient being informed and accepting to participate in the study with signature of informed consent
* HIV positive serology
* Clinical and radiological suspicion of cerebral toxoplasmosis justifying the start of specific antitoxoplasmic therapy

Exclusion Criteria:

* Protected patient
* Patient uncovered by social insurance
* Specific antitoxoplasmic therapy already initiated since 72h or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AIDS patients from the French West Indies and French Guiana having clinical and radiological suspicion of cerebral toxoplasmosis
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

SECONDARY OUTCOMES:
Isolation, genetic typing and storage of T. gondii strains collected among AIDS patients with cerebral toxoplasmosis from the DFA. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel AJZENBERG, PharmD, PhD, Study Director — CHU Limoges
Locations (5):
- France (5):
  - Service des Maladies Infectieuses - CHU de Pointe à Pitre, Pointe à Pitre, Guadeloupe
  - Dermatologie et CISIH- CH Andrée Rosemon, Guyane-Française, Guyane-Française
  - Médecine- CH Ouest Guyanais, Guyane-Français, Guyane-Français
  - Services Maladies Infectieuses et Tropicales- CHU Fort-de-France, Fort-de-France
  - Maladies Infectieuses et Tropicales - CH Andrée Rosemon, Guyane-Française

REFERENCES:
- [Result] Ajzenberg D, Lamaury I, Demar M, Vautrin C, Cabie A, Simon S, Nicolas M, Desbois-Nogard N, Boukhari R, Riahi H, Darde ML, Massip P, Dupon M, Preux PM, Labrunie A, Boncoeur MP. Performance Testing of PCR Assay in Blood Samples for the Diagnosis of Toxoplasmic Encephalitis in AIDS Patients from the French Departments of America and Genetic Diversity of Toxoplasma gondii: A Prospective and Multicentric Study. PLoS Negl Trop Dis. 2016 Jun 29;10(6):e0004790. doi: 10.1371/journal.pntd.0004790. eCollection 2016 Jun. PMID 27355620